CLINICAL TRIAL: NCT00548990
Title: Physical Activity, Aging and Immune Function
Brief Title: The Immune Function Intervention Trial
Acronym: ImFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0088; NIH R01 AG-18861
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Immune Response
MeSH Terms: interventions — Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): a 10-month moderate aerobic exercise training program
  Interventions: Behavioral: cardiovascular exercise training
- 2 (Placebo Comparator): flexibility/balance control group
  Interventions: Behavioral: flexibility/balance control

INTERVENTIONS:
Behavioral: cardiovascular exercise training
  Arms: 1
Behavioral: flexibility/balance control
  Arms: 2

SUMMARY:
The purpose of the study is to examine whether cardiovascular exercise training improves immune responses to vaccination in previously sedentary older adults.

DETAILED DESCRIPTION:
The extent to which exercise training or long-term physical activity influences poorly regulated immune function in the elderly is unclear. Preliminary evidence suggests that exercise training may improve various immune function measures in older adults. Although such findings have the potential to be of substantial public health importance, the majority of studies have suffered from small sample sizes, inadequate measurement of physical fitness, and weak research designs.

This study is designed to overcome these limitations by employing a longitudinal randomized controlled trial examining the effect of exercise training on clinically relevant immune function measures in older adults (65-80 years). Moreover, relationships between several factors known to be altered by exercise training and changes in immune function will be assessed. As such, there are two specific aims to be addressed. In Aim 1, a 10-month exercise trial will determine whether moderate intensity aerobic exercise training can improve immune function in previously sedentary older adults. In Aim 2, the role played by physiological, behavioral, and psychosocial factors in the relationship between exercise training and improved immune function will be examined.

150 sedentary participants will be randomly assigned to either a 10-month moderate aerobic exercise training program or a sedentary control group. Clinically relevant measures of immune function including the delayed-type hypersensitivity (DTH) response to a battery of antigens and the antibody response to tetanus toxoid and influenza virus vaccination will be assessed before, during and after the intervention. We hypothesize that exercise training will result in improved immune responses including higher peak antibody titers and DTH responses, and sustained levels of protective antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Ages 62-82
* Ability to participate in an exercise program
* Medical clearance by primary physician
* Non-smoker
* BMI 22-38
* Independently living
* Post-menopausal
* Sedentary for over 6 months

Exclusion Criteria:

* No recent history (within 6 months) of infection or vaccination
* History of systemic reactions to vaccination
* History of cancer
* Severe allergies/asthma requiring prescription medication
* Splenectomy or transplant patient
* Chronic Obstructive Pulmonary Disease (COPD)
* HIV positive
* Uncontrolled diabetes or hypertension
* Severe arthritis
* Mental illness or clinical depression
* Impaired cognitive status

Ages: 62 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
antibody responses to influenza and tetanus toxoid vaccination and delayed type hypersensitivity responses to fungal antigens | baseline, 6 and 10 months

SECONDARY OUTCOMES:
cardiovascular fitness
psychosocial outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Woods, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Background] Woods JA, Lowder TW, Keylock KT. Can exercise training improve immune function in the aged? Ann N Y Acad Sci. 2002 Apr;959:117-27. doi: 10.1111/j.1749-6632.2002.tb02088.x. PMID 11976191
- [Background] Woods JA, Ceddia MA, Wolters BW, Evans JK, Lu Q, McAuley E. Effects of 6 months of moderate aerobic exercise training on immune function in the elderly. Mech Ageing Dev. 1999 Jun 1;109(1):1-19. doi: 10.1016/s0047-6374(99)00014-7. PMID 10405985
- [Background] Kohut ML, Cooper MM, Nickolaus MS, Russell DR, Cunnick JE. Exercise and psychosocial factors modulate immunity to influenza vaccine in elderly individuals. J Gerontol A Biol Sci Med Sci. 2002 Sep;57(9):M557-62. doi: 10.1093/gerona/57.9.m557. PMID 12196490